CLINICAL TRIAL: NCT00215384
Title: Study in Patients With COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dey (Industry)
Responsible Party: Director, Clinical Affairs, Dey
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DL-052
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2010-11-11 (Estimated); Status verified 2008-02

CONDITIONS: COPD
Keywords: COPD; formoterol
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Formoterol Fumarate

INTERVENTIONS:
Drug: Formoterol Fumarate

SUMMARY:
The purpose of this study is to determine which dose of the investigational drug is the most safe and effective compared to the control drug.

ELIGIBILITY:
Inclusion Criteria:

-History of COPD and cigarette smoking

Exclusion Criteria:

* Clinical diagnosis of asthma.
* Chest X-ray that is diagnostic of a significant pulmonary disease other than COPD
* Disease of other major organ systems

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35
Dates: Primary Completion 2003-04 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome variable is the measure of lung function.

SECONDARY OUTCOMES:
Change in lung function will be examined as a secondary outcome, as well as vital signs, physical examination, adverse even reporting, etc.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Research Site, Los Angeles, California
  - Research Site, Upland, California
  - Research Site, Denver, Colorado
  - Research Site, Hines, Illinois
  - Research Site, Missoula, Montana
  - Research Site, Medford, Oregon
  - Research Site, Tacoma, Washington